CLINICAL TRIAL: NCT04917003
Title: Safety and Efficacy of Remote Ischemic Conditioning Combined Encephaloduroarteriosynangiosis（EDAS）on Ischemic Moyamoya Disease: A Prospective, Randomized, Controlled Study
Brief Title: Safety and Efficacy of Remote Ischemic Conditioning Combined EDAS on Ischemic Moyamoya Disease
Acronym: RIC-IMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIC-IMD
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Moyamoya Disease
Keywords: moyamoya disease; EDAS; remote ischemic conditioning; cerebral blood flow
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): Patients who are allocated into RIC group will undergo the first EDAS surgery combined 3-month remote ischemic conditioning (RIC) treatment. The opposite operation will be performed at 3 months after the first operation.
  RIC is a non-invasive therapy that performed by an electric auto-control device with cuff placed on arm. RIC procedures consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on one arm.
  EDAS involves placement of an external carotid artery branch beneath the dura in the ischemic territories. The superficial temporal artery (STA) was commonly used.
  Interventions: Other: RIC plus EDAS
- control group (Other): Patients who are allocated into the control group will accept EDAS surgery twice. The second operation will be performed at 3 months after the first operation.
  EDAS involves placement of an external carotid artery branch beneath the dura in the ischemic territories. The superficial temporal artery (STA) was commonly used. Under certain circumstances, depending on the territory at risk, the occipital artery was also used. The donor vessel with the strip of galea (the arterial bridge) was detached from the pericranium or the fascia below, and two burr holes are made beneath the proximal and distal ends of the arterial bridge. The burr holes, with an average size of 3.0 × 8.0 cm, were connected by mill to make an oval bone flap and the dura was exposed. The target artery was then sewn to the dura using 10-0 Prolene suture. The bone flap was closed after cutting out the entry and exit sites for the target artery.
  Interventions: Other: EDAS

INTERVENTIONS:
Other: RIC plus EDAS — Patients who are allocated into RIC group will undergo EDAS surgery combined 3-month RIC treatment. The opposite operation will be performed at 3 months after the first operation.
  Arms: RIC group
Other: EDAS — Patients who are allocated into the control group will accept EDAS surgery twice. The second operation will be performed at 3 months after the first operation.
  Arms: control group

SUMMARY:
Encephaloduroarteriosynangiosis (EDAS) is widely used as an indirect technique for treatment of moyamoya disease. Nevertheless, this indirect surgery tends to establish insufficient collateral circulation in most adult MMD patients. Nowadays, there is a lack of adjuvant therapies for improving collateral circulation induced by indirect revascularization. This study aims to explore whether remote ischemic conditioning can improve the collateral circulation after indirect revascularization.

DETAILED DESCRIPTION:
Encephaloduroarteriosynangiosis (EDAS) is widely used as an indirect technique for treatment of moyamoya disease. Nevertheless, this indirect surgery tends to establish insufficient collateral circulation in most adult MMD patients. Nowadays, there is a lack of adjuvant therapies for improving collateral circulation induced by indirect revascularization. Remote ischemic conditioning (RIC) is a noninvasive approach protecting the brain by inflating and deflating blood-pressure cuff placed on the upper limbs. It has been confirmed to improve cerebral perfusion by promoting angiogenesis and arteriogenesis in ischemic animal brain. In addition, daily remote ischemic conditioning is a promising technique to ameliorate chronic cerebrovascular disease like intracranial atherosclerotic stenosis, small-vessel disease.

Thus, this study aims to explore whether remote ischemic conditioning can improve the collateral circulation after indirect revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who were diagnosed as moyamoya disease by the diagnostic criteria recommended by the Research Committee on MMD of the Ministry of Health and Welfare of Japan in 2012.
2. Suzuki stage: 2-5 stage
3. Age: between 18 and 65 years old
4. Subjects present with ischemic stroke or transient ischemic attack.
5. Subjects who plan to accept the first EDAS surgery.
6. Informed consent obtained from patient or patient's surrogate

Exclusion Criteria:

1. Acute ischemic stroke occurred within one month.
2. Suffered Intracranial hemorrhage before
3. Subjects with large infarction spread widely over the territory of a main arterial trunk
4. Aneurysms in the main arterial trunk
5. Severe cardiac diseases like atrial fibrillation，valvular disease，heart failure, infective endocarditis and so on.
6. Malignant tumors or severe disordered function of the heart, lung, liver or kidney.
7. Severe hemostatic disorder or severe coagulation dysfunction.
8. Uncontrolled diabetes mellitus with a serum fasting blood glucose level>300 mg/dL, or requires insulin; hypertension with a systolic blood pressure over 180 mmHg or a diastolic blood pressure over 110 mmHg.
9. Severe injury on upper limbs.
10. Pregnant or lactating women.
11. Life expectancy is less than 3 years.
12. Patients who are not suitable for this trial considered by researchers for other reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
rCBF changed ratio at operative side | From baseline to 3 months.
  Cerebral blood flow will be evaluated by dynamic susceptibility contrast-MRI examination，and relative cerebral blood flow(rCBF) changed ratio will be calculated by the formula: (rCBF in MCA territory/rCBF in cerebellum after treatment - rCBF in MCA territory/rCBF in cerebellum before treatment )/ rCBF in MCA territory/rCBF in cerebellum before treatment (the operative side). The higher value of rCBF improvement ratio means better imaging outcome.

SECONDARY OUTCOMES:
the change of TTP delay at operative side | From baseline to 3 months.
  Time to peak(TTP) will be evaluated by dynamic susceptibility contrast-MRI examination. The improvement of TTP delay at operative side will be calculated by the formula: the change of TTP delay =TTP delay in MCA territory before treatment - TTP delay in MCA territory after treatment (the operative side). The higher value means better imaging outcome.
rCBF changed ratio at non-operative side | From baseline to 3 months.
  Cerebral blood flow will be evaluated by dynamic susceptibility contrast-MRI examination，and relative cerebral blood flow(rCBF) changed ratio will be calculated by the formula: (rCBF in MCA territory/rCBF in cerebellum after treatment - rCBF in MCA territory/rCBF in cerebellum before treatment )/ rCBF in MCA territory/rCBF in cerebellum before treatment (the non-operative side). The higher value of rCBF improvement ratio means better imaging outcome.
the change of TTP delay at non-operative side | From baseline to 3 months.
  Time to peak(TTP) will be evaluated by dynamic susceptibility contrast-MRI examination. The improvement of TTP delay at non-operative side will be calculated by the formula: Improvement of TTP delay =TTP delay in MCA territory before treatment - TTP delay in MCA territory after treatment (the non-operative side). The higher value means better imaging outcome.
Incidence of major adverse cerebral event ( MACE) | From baseline to 3 months.
  MACE contains ischemic or hemorrhagic stroke, crescendo TIAs evaluated by registered Neurologists.
The change of luminal area of superficial temporal artery | From baseline to 3 months.
  The luminal area of STA can reflect the angiogenesis induced by EDAS to some extent, and it will be measured by TOF-MRA.
The degree of the collaterals from superficial temporal artery | From baseline to 3 months.
  The degree of the collaterals from superficial temporal artery will be evaluated by Transcranial Doppler ultrasound performed by an experienced technician. 0 for no collaterals from STA, 1 for little collaterals from STA, 2 for good collaterals from STA .
Volume of regions with hyperintense signal | From baseline to 3 months.
  Volume of regions with hyperintense signal where the maximum dimension should be larger than 8mm will be measured at axial T2, fluid-attenuated inversion recovery.
Number of regions with hyperintense signal | From baseline to 3 months.
  Number of regions with hyperintense signal will be counted at axial T2, fluid-attenuated inversion recovery.
RIC related Adverse events | From baseline to 3 months.
  Adverse events related to RIC treatment, such as local edema, erythema, skin lesions of the arms.
Flow velocity of superficial temporal artery at operative side | From baseline to 3 months.
  Flow velocity of superficial temporal artery at operative side will be evaluated by Transcranial Doppler ultrasound performed by an experienced technician.

CONTACTS AND LOCATIONS:
Locations (1):
- The 307th Hospital of the Chinese People's Liberation Army, Beijing, China